CLINICAL TRIAL: NCT02105012
Title: Randomized, Double-Blind, Chronic Dosing (4 Weeks), Four-Period, Five-Treatment, Incomplete Block, Cross-Over, Multi-Center Study to Assess the Efficacy and Safety of Four Doses of Budesonide Inhalation Aerosol (BD MDI, PT008) Relative to Placebo MDI in Adult Subjects With Mild to Moderate Persistent Asthma
Brief Title: Study to Assess the Efficacy and Safety of Budesonide (PT008) in Adult Subjects With Mild to Moderate Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PT008001
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Mild; moderate persistent; Adult
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BD MDI 320 µg (Experimental): Budesonide metered dose inhaler (BD MDI) 320 µg (PT008) administered as 2 inhalations BID
  Interventions: Drug: BD MDI 320 µg
- BD MDI 160 µg (Experimental): BD MDI 160 µg (PT008) administered as 2 inhalations BID
  Interventions: Drug: BD MDI 160 µg
- BD MDI 80 µg (Experimental): BD MDI 80 µg (PT008) administered as 2 inhalations BID
  Interventions: Drug: BD MDI 80 µg
- BD MDI 40 µg (Experimental): BD MDI 40 µg (PT008) administered as 2 inhalations BID
  Interventions: Drug: BD MDI 40 µg
- Placebo MDI (Placebo Comparator): Placebo MDI administered as 2 inhalations BID
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: BD MDI 320 µg — Budesonide Inhalation Aerosol administered as 2 inhalations BID
  Other Names: PT008
  Arms: BD MDI 320 µg
Drug: BD MDI 160 µg — Budesonide Inhalation Aerosol administered as 2 inhalations BID
  Other Names: PT008
  Arms: BD MDI 160 µg
Drug: BD MDI 80 µg — Budesonide Inhalation Aerosol administered as 2 inhalations BID
  Other Names: PT008
  Arms: BD MDI 80 µg
Drug: BD MDI 40 µg — Budesonide Inhalation Aerosol administered as 2 inhalations BID
  Other Names: PT008
  Arms: BD MDI 40 µg
Drug: Placebo MDI — Placebo MDI administered as 2 inhalations BID
  Arms: Placebo MDI

SUMMARY:
Study to assess the efficacy and safety of four doses of budesonide inhalation aerosol (BD MDI, PT008) relative to placebo MDI in adult subjects with mild to moderate persistent asthma.

DETAILED DESCRIPTION:
This is a randomized, double-blind, chronic dosing (4 weeks), four-period, five-treatment, incomplete block, cross-over, multicenter study to assess the efficacy and safety of four doses of budesonide inhalation aerosol (BD MDI, PT008) relative to placebo MDI in adult subjects with mild to moderate persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 - 65 years of age
* Diagnosis of mild to moderate persistent asthma, diagnosed at least 6 months prior to screening
* Currently receiving treatment with a low to medium dose of an inhaled corticosteroid (ICS) OR a combination of controller medications for at least 4 weeks preceding screening
* Pre-albuterol FEV1 of > 60% and < 85% of predicted normal value
* Reversibility: Increase in FEV1 of ≥ 12% and ≥ 200 mL over the pre-albuterol FEV1 within 30 - 60 minutes after the inhalation of 4 puffs of Ventolin hydrofluoroalkane (HFA)
* Asthma Symptom Criteria: Have required albuterol use on at least two of the last seven days and have an Asthma Control Questionnaire (ACQ) total score ≥ 1.5 prior to Randomization

Exclusion Criteria:

* Life-Threatening Asthma: A subject must not have life-threatening asthma defined as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s) within the 12 months prior to screening
* Worsening of Asthma: A subject must not have experienced a worsening of asthma which involved an emergency department visit, hospitalization or use of oral/parenteral corticosteroids within 6 weeks of screening
* Intermittent, Seasonal, or Exercise-Induced Asthma Alone: Subjects with only intermittent, seasonal or exercise-induced asthma are excluded from participation in this study
* Concurrent Respiratory Disease
* Pregnant women or nursing mothers
* A current diagnosis of Chronic Obstructive Pulmonary Disease (COPD
* Current smokers or subjects with a > 10 pack year history of cigarettes, cigars, or pipe smoking
* Respiratory tract infection within 6 weeks prior to Visit 1
* Subjects with documented myocardial infarction within a year from screening visit
* Clinically significant abnormal ECG
* Abnormal liver function tests defined as aspartate aminotransferase (AST), alanine aminotransferace (ALT), alkaline phosphatase or total bilirubin ≥ 1.5 times upper limit of normal on repeat testing
* Subjects who have cancer that has not been in complete remission for at least 5 years
* Drug Allergy: Subjects who have a history of hypersensitivity to any component of the metered-dose inhaler (MDI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dorinsky, MD, FCCP, Study Director — Pearl Therapeutics, Inc.
Locations (41):
- United States (41):
  - Pearl Therapeutics Study Site, Athens, Alabama
  - Pearl Therapeutics Study Site, Birmingham, Alabama
  - Pearl Therapeutics Study Site, Foley, Alabama
  - Pearl Therapeutics Study Site, Los Angeles, California
  - Pearl Therapeutics, Los Angeles, California
  - Pearl Therapeutics Study Site, Rolling Hills Estates, California
  - Pearl Therapeutics Study Site, San Diego, California
  - Pearl Therapeutics Study Site, Stockton, California
  - Pearl Therapeutics Study Site, Clearwater, Florida
  - Pearl Therapeutics Study Site, Clermont, Florida
  - Pearl Therapeutics Study Site, Miami, Florida
  - Pearl Therapeutics Study Site, Orlando, Florida
  - Pearl Therapeutics Study Site, Ormond Beach, Florida
  - Pearl Therapeutics Study Site, Saint Cloud, Florida
  - Pearl Therapeutics Study Site, Sebring, Florida
  - Pearl Therapeutics Study Site, Tampa, Florida
  - Pearl Therapeutics Study Site, Blue Island, Illinois
  - Pearl Therapeutics Study Site, North Dartmouth, Massachusetts
  - Pearl Therapeutics Study Site, Hazelwood, Missouri
  - Pearl Therapeutics Study Site, Skillman, New Jersey
  - Pearl Therapeutics Study Site, Charlotte, North Carolina
  - Pearl Therapeutics Study Site, Winston-Salem, North Carolina
  - Pearl Therapeutics Study Site, Cincinnati, Ohio
  - Pearl Therapeutics Study Site, Columbus, Ohio
  - Pearl Therapeutics Study Site, Dayton, Ohio
  - Pearl Therapeutics Study Site, Middleburg Heights, Ohio
  - Pearl Therapeutics Study Site, Oregon, Ohio
  - Pearl Therapeutics Study Site, Sylvania, Ohio
  - Pearl Therapeutics Study Site, Toledo, Ohio
  - Pearl Therapeutics Study Site, Oklahoma City, Oklahoma
  - Pearl Therapeutics Study Site, Lake Oswego, Oregon
  - Pearl Therapeutics Study Site, Medford, Oregon
  - Pearl Therapeutics Study Site, Greenville, South Carolina
  - Pearl Therapeutics Study Site, Spartanburg, South Carolina
  - Pearl Therapeutics Study Site, Rapid City, South Dakota
  - Pearl Therapeutics Study Site, Tullahoma, Tennessee
  - Pearl Therapeutics Study Site, El Paso, Texas
  - Pearl Therapeutics Study Site, Houston, Texas
  - Pearl Therapeutics Study Site, Plano, Texas
  - Pearl Therapeutics Study Site, San Antonio, Texas
  - Pearl Therapeutics Study Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 44 sites in the US from May 2015 to September 2015. Study participation maximum of 32 weeks.
Pre-assignment Details: A Randomized, Double-Blind, Chronic Dosing (4 Weeks), Four-Period, Five-Treatment, Incomplete Block, Cross-Over, Multi-Center Study to Assess the Efficacy and Safety of Four Doses of Budesonide Inhalation Aerosol (BD MDI, PT008) Relative to Placebo MDI in Adult Subjects With Mild to Moderate Persistent Asthma
Period: Overall Study
Arm/Group | All Subjects
Started | 147
BD MDI 320 µg | 124
BD MDI 160 µg | 132
BD MDI 80 µg | 64
BD MDI 40 µg | 63
Placebo MDI | 127
Completed | 114
Not Completed | 33
Not completed — Withdrawal by Subject | 11
Not completed — Protocol Specified Criteria | 9
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 4
Not completed — Physician Decision | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | All Subjects
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose Trough Forced Expiratory Volume in 1 Second (FEV1) at the End of the Treatment Period
Description: Change from baseline in morning pre-dose trough Forced Expiratory Volume in 1 second (FEV1) at the end of the Treatment Period.
Time Frame: Baseline to End of Treatment Period (Day 29 or Day 15 if Day 29 is missing)
Population: Modified Intent to Treat Population (MITT)
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- BD MDI 320 µg: Budesonide (BD) Metered Dose Inhaler (MDI) 320 µg
- BD MDI 160 µg: Budesonide (BD) Metered Dose Inhaler (MDI) 160 µg
- BD MDI 80 µg: Budesonide (BD) Metered Dose Inhaler (MDI) 80 µg
- BD MDI 40 µg: Budesonide (BD) Metered Dose Inhaler (MDI) 40 µg
- Placebo MDI: Placebo MDI.
Arm/Group | BD MDI 320 µg | BD MDI 160 µg | BD MDI 80 µg | BD MDI 40 µg | Placebo MDI
Number analyzed (Participants) | 109 | 109 | 56 | 56 | 111
Liters | -0.002 [-0.036 to 0.033] | -0.001 [-0.035 to 0.033] | -0.034 [-0.081 to 0.014] | -0.031 [-0.079 to 0.016] | -0.116 [-0.150 to -0.082]

2. Secondary Outcome: Change From Baseline in Mean Morning Pre-dose Diary Peak Expiratory Flow Rate (PEFR)
Description: Change From Baseline in Mean Morning Pre-dose Diary Peak Expiratory Flow Rate (PEFR)
Time Frame: Baseline to Last 7 Days of Treatment Period
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/min
Arm/Group | BD MDI 320 µg | BD MDI 160 µg | BD MDI 80 µg | BD MDI 40 µg | Placebo MDI
Number analyzed (Participants) | 105 | 107 | 55 | 50 | 107
Liters/min | -5.802 [-17.937 to 6.333] | -7.461 [-19.536 to 4.614] | -9.992 [-24.293 to 4.309] | -5.653 [-20.320 to 9.014] | -29.933 [-42.019 to -17.847]

3. Secondary Outcome: Change From Baseline in Mean Evening Pre-dose Diary Peak Expiratory Flow Rate (PEFR)
Description: Change From Baseline in Mean Evening Pre-dose Diary Peak Expiratory Flow Rate (PEFR)
Time Frame: Baseline to Last 7 Days of Treatment Period
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/min
Arm/Group | BD MDI 320 µg | BD MDI 160 µg | BD MDI 80 µg | BD MDI 40 µg | Placebo MDI
Number analyzed (Participants) | 105 | 108 | 52 | 52 | 110
Liters/min | -7.345 [-18.394 to 3.703] | -11.791 [-22.737 to -0.844] | -14.403 [-28.118 to -0.688] | -1.896 [-15.585 to 11.793] | -32.807 [-43.712 to -21.902]

4. Secondary Outcome: Change From Baseline in Mean Number of Puffs of Rescue Ventolin HFA
Description: Change from baseline in mean number of puffs of rescue Ventolin HFA
Time Frame: Baseline to Last 7 Days of Treatment
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs/Day
Arm/Group | BD MDI 320 µg | BD MDI 160 µg | BD MDI 80 µg | BD MDI 40 µg | Placebo MDI
Number analyzed (Participants) | 111 | 115 | 56 | 56 | 114
Puffs/Day | -0.140 [-0.531 to 0.251] | -0.268 [-0.654 to 0.119] | -0.312 [-0.810 to 0.186] | -0.095 [-0.592 to 0.402] | 0.606 [0.218 to 0.994]

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score
Description: The ACQ-5 measures 5 symptoms (woken at night by symptoms, wake in the morning with symptoms, limitation of daily activities, shortness of breath, and wheeze). The scale is 0-6, where 0=minimum and 6=maximum
Time Frame: Baseline to End of Treatment Period (Day 29 or Day 15 if Day 29 is missing)
Population: MITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | BD MDI 320 µg | BD MDI 160 µg | BD MDI 80 µg | BD MDI 40 µg | Placebo MDI
Number analyzed (Participants) | 109 | 114 | 57 | 57 | 115
Scores on a scale | -0.575 [-0.730 to -0.420] | -0.565 [-0.717 to -0.412] | -0.515 [-0.714 to -0.317] | -0.407 [-0.605 to -0.209] | -0.100 [-0.252 to 0.052]

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time subjects received their first dose of study medication, during the entire study period, and up to 14 days from the date of the last study medication dose.
Description: The Safety population was defined as all subjects who were randomized to treatment and received at least 1 dose of the study treatment. Subjects in the Safety population were analyzed according to the treatment received.
Arm/Group | BD MDI 320 µg | BD MDI 160 µg | BD MDI 80 µg | BD MDI 40 µg | Placebo MDI
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/132 | 2/64 | 0/63 | 0/127
Other Adverse Events (participants affected / at risk) | 7/124 | 7/132 | 1/64 | 2/63 | 12/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BD MDI 320 µg (N=124) | BD MDI 160 µg (N=132) | BD MDI 80 µg (N=64) | BD MDI 40 µg (N=63) | Placebo MDI (N=127)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BD MDI 320 µg (N=124) | BD MDI 160 µg (N=132) | BD MDI 80 µg (N=64) | BD MDI 40 µg (N=63) | Placebo MDI (N=127)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.